CLINICAL TRIAL: NCT00398775
Title: Procalcitonin Guided Antimicrobial Discontinuation in Hospitalised Patients With Fever of Unknown Etiology
Brief Title: Procalcitonin in Fever of Unknown Etiology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low recruitment
Sponsor: Changi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/36
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Fever
Keywords: procalcitonin guided antibiotic discontinuation; fever of unknown origin
MeSH Terms: conditions — Fever; Fever of Unknown Origin

INTERVENTIONS:
Procedure: antibiotic discontinuation

SUMMARY:
The purpose of this study is to determine whether new blood test (procalcitonin) can help to reduce unnecessary use of antibiotics in patients with unexplained fever.

Although fever is most commonly caused by bacterial infection there are multiple other conditions that can cause fever. It can be caused by viral infection. It can also be caused by other non infectious disease. Patients with malignancy, inflammation (such as gout or arthritis), or clots in veins can present with fever. Occasionally medications themselves can cause fever. If fever is not caused by infection antibiotics will not help. Instead they may cause side effects such as diarrhea and allergic reactions. We want to determine whether simple blood test (procalcitonin) can help us to make a difference between fever caused by infection and fever caused by others (above mentioned) non-infectious problems. We also want to determine whether such test would help us to reduce unnecessary antibiotic use and help us to find faster the real cause of the fever.

A total of 90 patients with the unexplained fever will be participating in this study. This study will involve single, additional blood test, performed only if patient continue to have fever despite a few days of investigations and therapy with antibiotics.

Patients will be assigned by drawing to one of two groups. In the first group blood test (procalcitonin) will help a doctor to decide whether to stop or continue antibiotics. If procalcitonin level is high antibiotics will be continued and the doctor will most probably order additional tests to determine the source of infection. If procalcitonin level is low serious bacterial infection is unlikely. The antibiotics will be stopped and a doctor will try to look for other cause of fever.

In the second group blood for the tests will be collected but not reported to a doctor. You will be treated in traditional manner by a doctor.

By following this procedure we will be able to determine whether therapy guided by procalcitonin level is as safe and possibly more effective than traditional approach. This study does not involve any other tests or study medications. We will attempt to contact all patients one month later by phone to determine whether you remain well after discharge.

DETAILED DESCRIPTION:
Antimicrobial resistance has increasingly become a threat to patient safety in health care settings.1 Several studies have identified the inappropriate use of antimicrobials as important risk factor for antimicrobial resistance and the important area of opportunity for increasing patient safety and improving patient outcomes.2 High rates of antimicrobial use have been linked to high rates of antimicrobial resistance,3 and increased exposure to antimicrobials has been associated with an increased probability of colonization with resistant pathogens. It has also been shown that antimicrobial control results in significant cost savings4 and it may reduce antimicrobial resistance Surveys reveal that 25 - 33% of hospitalized patients receive antibiotics6 and that 22 - 65% of antibiotic use in hospitalized patients is inappropriate.7

Reasons for inappropriate antimicrobial therapy include:

1. treating anybody with fever (even when it is not caused by infection) with broad spectrum antibiotics
2. treating colonization or contamination (rather than real infection)
3. continuing antibiotics even when infection was cured or is unlikely8

It is quite clear that clinicians need reliable marker for bacterial infections that would allow an early diagnosis, inform about the course and prognosis of the disease and facilitate therapeutic decisions.9 Procalcitonin covers these features better as compared to other, more commonly used biomarkers (such as CRP).10 It has been shown recently that procalcitonin guidance substantially reduces antibiotic use in community-acquired pneumonia without compromising patients' safety. 11, 12 However, the efficacy and safety of PGAD in hospitalized patients with undefined fever has not been previously investigated.

We think that PGAD should be equally safe and effective intervention in hospitalized patients with fever of unknown etiology. It should help to reduce inappropriate antibiotic use and in effect, help to control antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

1. All hospitalized patients admitted to general medical or GRM wards with fever and no obvious source of infection, and
2. remain febrile after 72 hours of empiric, antimicrobial therapy, and
3. initial blood cultures are negative.

Exclusion Criteria:

1. Patients with clinically suspected infection (strongly suggestive symptoms, signs or laboratory/imaging studies) such as pneumonia, urinary tract infection, meningitis, endocarditis, skin and soft tissue infection, etc.
2. Confirmed bacterial, viral or fungal infection (positive stain, culture or serology from appropriate clinical specimen).
3. Hypotension (systolic blood pressure <90mmHg)
4. Respiratory failure (oxygen requirement > 4L/min via nasal canula)
5. Patients admitted to intensive care unit.
6. Severely immunocompromised patients: (febrile neutropenia, HIV infection with CD4 count < 200, immuno-suppressive therapy).
7. Patients younger than 21.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Exposure to systemic antimicrobial treatment:
duration of antibiotic treatment (in days).
total antibiotic exposure (in defined daily doses).

SECONDARY OUTCOMES:
28-day case-fatality rate (in %)
Length of hospital stay (in days)
Costs of antimicrobial therapy (in SGD)
Rate of nosocomial super-infection (in N super-infections per 100 patients)
Isolation of multi-resistant microorganisms (in clinical isolates per 100 patient-days)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej P Chlebicki, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Briel M, Christ-Crain M, Young J, Schuetz P, Huber P, Periat P, Bucher HC, Muller B. Procalcitonin-guided antibiotic use versus a standard approach for acute respiratory tract infections in primary care: study protocol for a randomised controlled trial and baseline characteristics of participating general practitioners [ISRCTN73182671]. BMC Fam Pract. 2005 Aug 18;6:34. doi: 10.1186/1471-2296-6-34. PMID 16107222
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Christ-Crain M, Muller B. Procalcitonin in bacterial infections--hype, hope, more or less? Swiss Med Wkly. 2005 Aug 6;135(31-32):451-60. doi: 10.4414/smw.2005.11169. PMID 16208582